CLINICAL TRIAL: NCT00356369
Title: Phase IIb Primary Vaccination Study to Evaluate Non-Inferiority & Persistence of the Immune Response of GSK Biologicals' MenACWY Conjugate Vaccine (Intramuscularly) vs Mencevax ACWY (Subcutaneously) to Healthy Subjects (11-55 Years of Age)
Brief Title: Study in Adolescents/Adults to Evaluate Non-inferiority&Persistence up to 5 Years of GSK Bio MenACWY Conjugate Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107386; 107392 (Ext: Y1) (Other: GSK); 107398 (Ext: Y2) (Other: GSK); 107402 (Ext: Y3) (Other: GSK); 107404 (Ext: Y4) (Other: GSK); 107406 (Ext: Y5) (Other: GSK); NCT00356499 (obsolete NCT alias); NCT00356538 (obsolete NCT alias); NCT00356577 (obsolete NCT alias); NCT00356694 (obsolete NCT alias); NCT00356876 (obsolete NCT alias)
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-05

CONDITIONS: Infections, Meningococcal
Keywords: Immunogenicity; Healthy; Persistence; Meningococcal vaccine; Non-inferiority; Meningococcal A C W Y Diseases; meningococcal serogroups A, C, W & Y diseases
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines

ARMS (2):
- Nimenrix Group (Experimental): Subjects receiving GSK Biologicals' meningococcal vaccine 134612
  Interventions: Biological: meningococcal ACWY (vaccine)
- Mencevax Group (Active Comparator): Subjects receiving Mencevax™ ACWY
  Interventions: Biological: Mencevax™ ACWY

INTERVENTIONS:
Biological: meningococcal ACWY (vaccine) — One intramuscular dose.
  Arms: Nimenrix Group
Biological: Mencevax™ ACWY — One subcutaneous dose.
  Arms: Mencevax Group

SUMMARY:
Meningococcal disease is mostly caused by N. meningitidis of serogroups A, B, C, W-135, Y. Meningococcal polysaccharide-conjugate vaccines have the advantage to induce a T-cell dependant immune response while the existing polysaccharide vaccines induce a T-cell independent response, i.e. with no immune memory response. GSK Biologicals has developed a combined Men ACWY conjugate vaccine intended to protect against meningococcal disease due to serogroups A, C, W-135 and Y. In the vaccination phase of this study, the new MenACWY-TT conjugate vaccine will be evaluated in adolescents and adults using Mencevax™ ACWY as control. In the long-term follow-up phase (extension phase) of the study, the long-term protection offered by the new MenACWY-TT conjugate vaccine will be assessed up to five years after the vaccination in adolescents and adults using Mencevax™ ACWY as control. This protocol posting deals with objectives & outcome measures of both the primary & extension phases.

DETAILED DESCRIPTION:
All subjects will have 7 blood samples taken: prior to and one month after vaccination and one, two, three, four and five years after vaccination. No new subjects will be enrolled in the extension phases of this Phase IIb study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, September 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents/ legally acceptable representative can and will comply with the requirements of the protocol.
* A male or female between, and including, 11 and 55 years of age at the time of vaccination.
* Written informed consent obtained from the subject/ from the parent or legally acceptable representative of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her knowledge and/or his/her parents/legally acceptable representative's knowledge.
* If the subject is female, she must be of non-childbearing potential; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, and must agree to continue such precautions for two months after completion of the vaccination series. Female subjects in childbearing potential who are not abstinent must have a negative pregnancy test.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine(s).
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C W and/or Y within the last five previous years.
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroup A, C W and/or Y.
* History of meningococcal disease due to serogroup A, C, W or Y.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* History of Guillain-Barré syndrome.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Specific criteria to be checked at each study visit for the long term follow-up:

* History of meningococcal serogroup A,C, W and Y disease.
* Administration of a meningococcal polysaccharide or a meningococcal polysaccharide conjugate vaccine not planned in the protocol.

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2006-12-23 (Actual); Primary Completion 2007-09-07 (Actual); Study Completion 2008-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Philippines (2):
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Manila
- GSK Investigational Site, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Borja-Tabora CF, Montalban C, Memish ZA, Boutriau D, Kolhe D, Miller JM, Van der Wielen M. Long-term immunogenicity and safety after a single dose of the quadrivalent meningococcal serogroups A, C, W, and Y tetanus toxoid conjugate vaccine in adolescents and adults: 5-year follow-up of an open, randomized trial. BMC Infect Dis. 2015 Oct 6;15:409. doi: 10.1186/s12879-015-1138-y. PMID 26437712
- [Derived] Borja-Tabora C, Montalban C, Memish ZA, Van der Wielen M, Bianco V, Boutriau D, Miller J. Immune response, antibody persistence, and safety of a single dose of the quadrivalent meningococcal serogroups A, C, W-135, and Y tetanus toxoid conjugate vaccine in adolescents and adults: results of an open, randomised, controlled study. BMC Infect Dis. 2013 Mar 5;13:116. doi: 10.1186/1471-2334-13-116. PMID 23510357
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 107386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Nimenrix Group: Subjects who received one dose of Nimenrix™ vaccine, administrated intramuscularly (IM) by injection in the non-dominant deltoid region.
- Mencevax Group: Subjects who received one dose of Mencevax™ ACWY vaccine, administrated subcutaneous by injection into the non-dominant upper arm.
Period: Active Phase
Arm/Group | Nimenrix Group | Mencevax Group
Started | 374 | 126
Completed | 372 | 125
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: Year 1
Arm/Group | Nimenrix Group | Mencevax Group
Started | 364 | 121
Completed | 364 | 121
Not Completed | 0 | 0
Period: Year 2
Arm/Group | Nimenrix Group | Mencevax Group
Started | 354 | 117
Completed | 354 | 117
Not Completed | 0 | 0
Period: Year 3
Arm/Group | Nimenrix Group | Mencevax Group
Started | 344 | 116
Completed | 344 | 116
Not Completed | 0 | 0
Period: Year 4
Arm/Group | Nimenrix Group | Mencevax Group
Started | 317 | 109
Completed | 317 | 109
Not Completed | 0 | 0
Period: Year 5
Arm/Group | Nimenrix Group | Mencevax Group
Started | 299 | 105
Completed | 299 | 105
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nimenrix Group: Subjects who received one dose of Nimenrix™ vaccine, administrated intramuscularly (IM) in the non-dominant deltoid region.
- Total: Total of all reporting groups
Arm/Group | Nimenrix Group | Mencevax Group | Total
Number analyzed (Participants) | 374 | 126 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.6 (7.62) | 19.3 (8.58) | 18.78 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 60 | 228
  Male | 206 | 66 | 272
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian-East Asian heritage | 1 | 0 | 1
  Geographic ancestry: Asian-South East Asian heritage | 298 | 101 | 399
  Geographic ancestry: White-Arabic/North African heritage | 75 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Response to Meningococcal Antigens for Serum Bactericidal Assay Using Rabbit Complement (rSBA)
Description: Response to vaccine antigen was defined as: for initially seronegative subjects [subjects with serum bactericidal assay using rabbit complement (rSBA) titer lower than (<) 1:8, post-vaccination rSBA titer greater than or equal to (≥) 1:32] and for initially seropositive (subjects with rSBA titer ≥ 1:8), at least 4-fold increase in rSBA titer from pre to post vaccination.
Time Frame: One month post vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 329 | 113
Percentage of subjects
  rSBA-MenA: number analyzed (Participants) | 289 | 99
  rSBA-MenA | 82.7 [77.8 to 86.9] | 69.7 [59.6 to 78.5]
  rSBA-MenC: number analyzed (Participants) | 324 | 113
  rSBA-MenC | 94.4 [91.4 to 96.7] | 90.3 [83.2 to 95]
  rSBA-MenW-135: number analyzed (Participants) | 326 | 109
  rSBA-MenW-135 | 96.3 [93.7 to 98.1] | 91.7 [84.9 to 96.2]
  rSBA-MenY | 93 [89.7 to 95.5] | 85 [77 to 91]
Statistical Analysis 1: Comparison: Nimenrix Group vs Mencevax Group; To evaluate the non-inferiority of the vaccine response* induced by the MenACWY-TT vaccine when compared to the licensed MenACWY vaccine; Test type: Non-Inferiority — Criterion indicative of non-inferiority: Lower limit of the standardized asymptotic 95% confidence interval (CI) for the difference between MenACWY-TT and (minus) MenACWY in the percentage of subjects with bactericidal vaccine response was greater than (>) -15%; Difference in % for rSBA-MenA antibodies = 13, 95% CI 2-sided [3.52 to 23.5]
Statistical Analysis 2: Comparison: Nimenrix Group vs Mencevax Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Criterion indicative of non-inferiority: Lower limit of the standardized asymptotic 95% confidence interval (CI) for the difference between MenACWY-TT and (minus) MenACWY in the percentage of subjects with bactericidal vaccine response was ≥ -12%; Difference in % for rSBA-MenC antibodies = 4.18, 95% CI 2-sided [-1.03 to 11.36]
Statistical Analysis 3: Comparison: Nimenrix Group vs Mencevax Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in%for rSBA-MenW-135 antibody = 4.58, 95% CI 2-sided [-0.07 to 11.49]
Statistical Analysis 4: Comparison: Nimenrix Group vs Mencevax Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in % for rSBA-MenY antibodies = 8.05, 95% CI 2-sided [1.72 to 16.17]

2. Primary Outcome: Occurrence of Any Grade 3 Systemic Symptoms
Description: Local symptom, Grade 3 = pain that prevented normal activity and redness/ swelling spreading beyond (>) 50 millimeters (mm).
  General symptom, Grade 3 = symptom that prevented normal activity and fever (orally) >39.5 °C.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects from whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 374 | 126
Participants
  Any Grade 3 unsolicited | 12 | 1
  Grade 3 solicited general | 5 | 0
  Grade 3 solicited local | 9 | 1
Statistical Analysis 1: Comparison: Nimenrix Group vs Mencevax Group; To evaluate the non-inferiority of the MenACWY-TT conjugate vaccine when compared to the licensed MenACWY vaccine in terms of the incidence of any Grade 3 systemic symptom within 4 days after vaccination; Test type: Non-Inferiority — Criterion indicative of non-inferiority: Upper limit of the standardized asymptotic 95% CI on the difference between MenACWY- TT and (minus) MenACWY in the incidence of Grade 3 systemic symptoms was below 5%; Difference in % Grade 3 general symptoms = 1.34, 95% CI 2-sided [-1.64 to 3.09]

3. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using Rabbit Complement Against Neisseria Meningitidis Serogroups A, C, W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8 and (≥) 1:128.
Time Frame: Prior to and 1 Month after vaccination
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects from whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 341 | 114
Participants
  rSBA-MenA (PRE) ≥ 1:8: number analyzed (Participants) | 305 | 101
  rSBA-MenA (PRE) ≥ 1:8 | 290 | 88
  rSBA-MenA (PI [M1]) ≥ 1:8: number analyzed (Participants) | 323 | 112
  rSBA-MenA (PI [M1]) ≥ 1:8 | 323 | 112
  rSBA-MenA (PRE) ≥ 1:128: number analyzed (Participants) | 305 | 101
  rSBA-MenA (PRE) ≥ 1:128 | 273 | 81
  rSBA-MenA (PI [M1]) ≥ 1:128: number analyzed (Participants) | 323 | 112
  rSBA-MenA (PI [M1]) ≥ 1:128 | 322 | 112
  rSBA-MenC (PRE) ≥ 1:8: number analyzed (Participants) | 324 | 113
  rSBA-MenC (PRE) ≥ 1:8 | 253 | 96
  rSBA-MenC (PI [M1]) ≥ 1:8 | 340 | 114
  rSBA-MenC (PRE) ≥ 1:128: number analyzed (Participants) | 324 | 113
  rSBA-MenC (PRE) ≥ 1:128 | 172 | 56
  rSBA-MenC (PI [M1]) ≥ 1:128 | 340 | 112
  rSBA-MenW-135 (PRE) ≥ 1:8: number analyzed (Participants) | 327 | 109
  rSBA-MenW-135 (PRE) ≥ 1:8 | 247 | 89
  rSBA-MenW-135 (PI [M1]) ≥ 1:8: number analyzed (Participants) | 340 | 114
  rSBA-MenW-135 (PI [M1]) ≥ 1:8 | 339 | 114
  rSBA-MenW-135 (PRE) ≥ 1:128: number analyzed (Participants) | 327 | 109
  rSBA-MenW-135 (PRE) ≥ 1:128 | 191 | 67
  rSBA-MenW-135 (PI [M1]) ≥ 1:128: number analyzed (Participants) | 340 | 114
  rSBA-MenW-135 (PI [M1]) ≥ 1:128 | 338 | 114
  rSBA-MenY (PRE) ≥ 1:8: number analyzed (Participants) | 330 | 113
  rSBA-MenY (PRE) ≥ 1:8 | 306 | 105
  rSBA-MenY (PI [M1]) ≥ 1:8: number analyzed (Participants) | 340 | 114
  rSBA-MenY (PI [M1]) ≥ 1:8 | 340 | 114
  rSBA-MenY (PRE) ≥ 1:128: number analyzed (Participants) | 330 | 113
  rSBA-MenY (PRE) ≥ 1:128 | 264 | 88
  rSBA-MenY (PI [M1]) ≥ 1:128: number analyzed (Participants) | 340 | 114
  rSBA-MenY (PI [M1]) ≥ 1:128 | 339 | 114

4. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as Geometric Mean Titers (GMTs).
Time Frame: Prior to and 1 Month after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 341 | 114
Titer
  rSBA-MenA (PRE): number analyzed (Participants) | 305 | 101
  rSBA-MenA (PRE) | 330.7 [285.8 to 382.7] | 227.8 [162.1 to 320.2]
  rSBA-MenA (PI [M1]): number analyzed (Participants) | 323 | 112
  rSBA-MenA (PI [M1]) | 4944.6 [4451.5 to 5492.5] | 2190.1 [1857.5 to 2582.2]
  rSBA-MenC (PRE): number analyzed (Participants) | 324 | 113
  rSBA-MenC (PRE) | 84.1 [68.5 to 103.4] | 114.1 [80.3 to 162]
  rSBA-MenC (PI [M1]) | 10073.7 [8699.9 to 11664.5] | 6545.6 [5047.5 to 8488.4]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 327 | 109
  rSBA-MenW-135 (PRE) | 93 [74.6 to 116] | 115.3 [81.6 to 162.9]
  rSBA-MenW-135 (PI [M1]): number analyzed (Participants) | 340 | 114
  rSBA-MenW-135 (PI [M1]) | 8576.5 [7614.9 to 9659.5] | 2969.5 [2439.4 to 3614.9]
  rSBA-MenY (PRE): number analyzed (Participants) | 330 | 113
  rSBA-MenY (PRE) | 310 [261.2 to 367.9] | 282.8 [209.9 to 380.8]
  rSBA-MenY (PI [M1]): number analyzed (Participants) | 340 | 114
  rSBA-MenY (PI [M1]) | 10315.2 [9317.1 to 11420.2] | 4573.7 [3863.9 to 5413.9]

5. Secondary Outcome: Number of Subjects With Anti-Polysaccharide (Anti-PS) Antibodies
Description: The cut-off value for the anti-PS concentration was greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL) and ≥ 2.0 μg/mL.
Time Frame: Prior to and 1 Month after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 341 | 114
Participants
  Anti-PSA (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 316 | 107
  Anti-PSA (PRE) ≥ 0.3 μg/mL | 255 | 90
  Anti-PSA (PI [M1]) ≥ 0.3 μg/mL: number analyzed (Participants) | 340 | 113
  Anti-PSA (PI [M1]) ≥ 0.3 μg/mL | 339 | 113
  Anti-PSA (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 316 | 107
  Anti-PSA (PRE) ≥ 2.0 μg/mL | 137 | 53
  Anti-PSA (PI [M1]) ≥ 2.0 μg/mL: number analyzed (Participants) | 340 | 113
  Anti-PSA (PI [M1]) ≥ 2.0 μg/mL | 339 | 113
  Anti-PSC (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 334 | 110
  Anti-PSC (PRE) ≥ 0.3 μg/mL | 71 | 27
  Anti-PSC (PI [M1]) ≥ 0.3 μg/mL | 340 | 114
  Anti-PSC (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 334 | 110
  Anti-PSC (PRE) ≥ 2.0 μg/mL | 30 | 16
  Anti-PSC (PI [M1]) ≥ 2.0 μg/mL | 333 | 113
  Anti-PSW-135 (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 332 | 106
  Anti-PSW-135 (PRE) ≥ 0.3 μg/mL | 41 | 17
  Anti-PSW-135 (PI [M1]) ≥ 0.3 μg/mL: number analyzed (Participants) | 339 | 114
  Anti-PSW-135 (PI [M1]) ≥ 0.3 μg/mL | 335 | 113
  Anti-PSW-135 (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 332 | 106
  Anti-PSW-135 (PRE) ≥ 2.0 μg/mL | 11 | 4
  Anti-PSW-135 (PI [M1]) ≥ 2.0 μg/mL: number analyzed (Participants) | 339 | 114
  Anti-PSW-135 (PI [M1]) ≥ 2.0 μg/mL | 314 | 106
  Anti-PSY (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 329 | 110
  Anti-PSY (PRE) ≥ 0.3 μg/mL | 55 | 23
  Anti-PSY (PI [M1]) ≥ 0.3 μg/mL: number analyzed (Participants) | 339 | 112
  Anti-PSY (PI [M1]) ≥ 0.3 μg/mL | 338 | 112
  Anti-PSY (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 329 | 110
  Anti-PSY (PRE) ≥ 2.0 μg/mL | 25 | 8
  Anti-PSY (PI [M1]) ≥ 2.0 μg/mL: number analyzed (Participants) | 339 | 112
  Anti-PSY (PI [M1]) ≥ 2.0 μg/mL | 328 | 109

6. Secondary Outcome: Concentration of Anti-PS Antibodies
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) and measured in micrograms/milliliter (µg/mL).
Time Frame: Prior to and 1 Month after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 341 | 114
μg/mL
  Anti-PSA (PRE): number analyzed (Participants) | 316 | 107
  Anti-PSA (PRE) | 1.4 [1.2 to 1.7] | 1.7 [1.3 to 2.3]
  Anti-PSA (PI [M1]): number analyzed (Participants) | 340 | 113
  Anti-PSA (PI [M1]) | 107.3 [92.7 to 124.1] | 53.6 [41.9 to 68.5]
  Anti-PSC (PRE): number analyzed (Participants) | 334 | 110
  Anti-PSC (PRE) | 0.3 [0.2 to 0.3] | 0.3 [0.2 to 0.4]
  Anti-PSC (PI [M1]) | 23.9 [21 to 27.2] | 43.9 [35.6 to 54.1]
  Anti-PSW-135 (PRE): number analyzed (Participants) | 332 | 106
  Anti-PSW-135 (PRE) | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.3]
  Anti-PSW-135 (PI [M1]): number analyzed (Participants) | 339 | 114
  Anti-PSW-135 (PI [M1]) | 18.6 [15.8 to 21.8] | 15.8 [12.1 to 20.7]
  Anti-PSY (PRE): number analyzed (Participants) | 329 | 110
  Anti-PSY (PRE) | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.3]
  Anti-PSY (PI [M1]): number analyzed (Participants) | 339 | 112
  Anti-PSY (PI [M1]) | 23.2 [19.9 to 26.9] | 23.6 [18.4 to 30.2]

7. Secondary Outcome: Number of Subjects With Anti-Tetanus (Anti-TT) Antibodies
Description: Cut-off values assessed were greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to and 1 Month after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 341 | 113
Participants
  Anti-TT (PRE): number analyzed (Participants) | 331 | 110
  Anti-TT (PRE) | 223 | 110
  Anti-TT (PI [M1]) | 326 | 113

8. Secondary Outcome: Concentration of Anti-TT Antibodies
Description: Concentrations are presented as geometric mean concentrations (GMCs) expressed in international units per milliliter (IU/mL).
Time Frame: Prior to and 1 Month after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 341 | 113
IU/mL
  Anti-TT (PRE): number analyzed (Participants) | 331 | 110
  Anti-TT (PRE) | 0.35 [0.29 to 0.43] | 0.28 [0.2 to 0.39]
  Anti-TT (PI [M1]) | 10.01 [8.34 to 12.03] | 0.27 [0.19 to 0.38]

9. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titres was greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: At Year 1
Population: The analysis was performed on the ATP cohort for persistence Year 1, which included all evaluable subjects who received the vaccine during the vaccination phase, without a previous dose of meningococcal serogroup A, C, W-135, or Y vaccines and who had available results for at least one tested antigen at the Year 1 time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 356 | 117
Participants
  rSBA-MenA (PI [M12]) ≥ 1:8: number analyzed (Participants) | 354 | 113
  rSBA-MenA (PI [M12]) ≥ 1:8 | 353 | 113
  rSBA-MenA (PI [M12]) ≥ 1:128: number analyzed (Participants) | 354 | 113
  rSBA-MenA (PI [M12]) ≥ 1:128 | 352 | 112
  rSBA-MenC (PI [M12]) ≥ 1:8: number analyzed (Participants) | 353 | 115
  rSBA-MenC (PI [M12]) ≥ 1:8 | 352 | 114
  rSBA-MenC (PI [M12]) ≥ 1:128: number analyzed (Participants) | 353 | 115
  rSBA-MenC (PI [M12]) ≥ 1:128 | 343 | 110
  rSBA-MenW-135 (PI [M12]) ≥ 1:8 | 355 | 117
  rSBA-MenW-135 (PI [M12]) ≥ 1:128 | 354 | 111
  rSBA-MenY (PI [M12]) ≥ 1:8: number analyzed (Participants) | 355 | 116
  rSBA-MenY (PI [M12]) ≥ 1:8 | 355 | 116
  rSBA-MenY (PI [M12]) ≥ 1:128: number analyzed (Participants) | 355 | 116
  rSBA-MenY (PI [M12]) ≥ 1:128 | 354 | 114

10. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as Geometric Mean Titers (GMTs).
Time Frame: At Year 1
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 356 | 117
Titer
  rSBA-MenA (PI [M12]): number analyzed (Participants) | 354 | 113
  rSBA-MenA (PI [M12]) | 2084.9 [1888.3 to 2302] | 1099.1 [931.6 to 1296.7]
  rSBA-MenC (PI [M12]): number analyzed (Participants) | 353 | 115
  rSBA-MenC (PI [M12]) | 1848.6 [1620.3 to 2109.2] | 1876.5 [1400.7 to 2514]
  rSBA-MenW-135 (PI [M12]) | 2993.5 [2618.8 to 3421.9] | 699.9 [569.3 to 860.4]
  rSBA-MenY (PI [M12]): number analyzed (Participants) | 355 | 116
  rSBA-MenY (PI [M12]) | 4207.1 [3767.3 to 4698.3] | 1386.5 [1104.2 to 1740.9]

11. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: At Year 2
Population: The analysis was performed on the ATP cohort for persistence Year 2, which included all evaluable subjects who received the vaccine during the vaccination phase, without a previous dose of meningococcal serogroup A, C, W-135, or Y vaccines and who had available results for at least one tested antigen at the Year 2 time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 346 | 112
Participants
  rSBA-MenA (PI [M24]) ≥ 1:8: number analyzed (Participants) | 338 | 102
  rSBA-MenA (PI [M24]) ≥ 1:8 | 337 | 101
  rSBA-MenA (PI [M24]) ≥ 1:128: number analyzed (Participants) | 338 | 102
  rSBA-MenA (PI [M24]) ≥ 1:128 | 335 | 98
  rSBA-MenC (PI [M24]) ≥ 1:8: number analyzed (Participants) | 345 | 112
  rSBA-MenC (PI [M24]) ≥ 1:8 | 343 | 110
  rSBA-MenC (PI [M24]) ≥ 1:128: number analyzed (Participants) | 345 | 112
  rSBA-MenC (PI [M24]) ≥ 1:128 | 332 | 103
  rSBA-MenW-135 (PI [M24]) ≥ 1:8: number analyzed (Participants) | 346 | 111
  rSBA-MenW-135 (PI [M24]) ≥ 1:8 | 344 | 100
  rSBA-MenW-135 (PI [M24]) ≥ 1:128: number analyzed (Participants) | 346 | 111
  rSBA-MenW-135 (PI [M24]) ≥ 1:128 | 341 | 90
  rSBA-MenY (PI [M24]) ≥ 1:8: number analyzed (Participants) | 345 | 111
  rSBA-MenY (PI [M24]) ≥ 1:8 | 344 | 110
  rSBA-MenY (PI [M24]) ≥ 1:128: number analyzed (Participants) | 345 | 111
  rSBA-MenY (PI [M24]) ≥ 1:128 | 342 | 105

12. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as Geometric Mean Titers (GMTs).
Time Frame: At Year 2
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Titre
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 346 | 112
Titre
  rSBA-MenA (PI [M24]): number analyzed (Participants) | 338 | 102
  rSBA-MenA (PI [M24]) | 1326.8 [1197.7 to 1469.7] | 698.9 [561.2 to 870.4]
  rSBA-MenC (PI [M24]): number analyzed (Participants) | 345 | 112
  rSBA-MenC (PI [M24]) | 1162 [1013.1 to 1332.9] | 1229.4 [876.4 to 1724.7]
  rSBA-MenW-135 (PI [M24]): number analyzed (Participants) | 346 | 111
  rSBA-MenW-135 (PI [M24]) | 1984.6 [1757.1 to 2241.4] | 319.1 [228 to 446.5]
  rSBA-MenY (PI [M24]): number analyzed (Participants) | 345 | 111
  rSBA-MenY (PI [M24]) | 3042.1 [2692.2 to 3437.5] | 850.2 [667.5 to 1082.9]

13. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: At Year 3
Population: The analysis was performed on the ATP cohort for persistence Year 3, which included all evaluable subjects who received the vaccine during the vaccination phase, without a previous dose of meningococcal serogroup A, C, W-135, or Y vaccines and who had available results for at least one tested antigen at the Year 3 time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 338 | 109
Participants
  rSBA-MenA (PI [M36]) ≥ 1:8: number analyzed (Participants) | 322 | 104
  rSBA-MenA (PI [M36]) ≥ 1:8 | 322 | 104
  rSBA-MenA (PI [M36]) ≥ 1:128: number analyzed (Participants) | 322 | 104
  rSBA-MenA (PI [M36]) ≥ 1:128 | 319 | 98
  rSBA-MenC (PI [M36]) ≥ 1:8: number analyzed (Participants) | 337 | 109
  rSBA-MenC (PI [M36]) ≥ 1:8 | 334 | 108
  rSBA-MenC (PI [M36]) ≥ 1:128: number analyzed (Participants) | 337 | 109
  rSBA-MenC (PI [M36]) ≥ 1:128 | 313 | 102
  rSBA-MenW-135 (PI [M36]) ≥ 1:8: number analyzed (Participants) | 336 | 105
  rSBA-MenW-135 (PI [M36]) ≥ 1:8 | 335 | 91
  rSBA-MenW-135 (PI [M36]) ≥ 1:128: number analyzed (Participants) | 336 | 105
  rSBA-MenW-135 (PI [M36]) ≥ 1:128 | 332 | 84
  rSBA-MenY (PI [M36]) ≥ 1:8: number analyzed (Participants) | 338 | 108
  rSBA-MenY (PI [M36]) ≥ 1:8 | 337 | 107
  rSBA-MenY (PI [M36]) ≥ 1:128: number analyzed (Participants) | 338 | 108
  rSBA-MenY (PI [M36]) ≥ 1:128 | 336 | 105

14. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as Geometric Mean Titers (GMTs).
Time Frame: At Year 3
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 338 | 109
Titer
  rSBA-MenA (PI [M36]): number analyzed (Participants) | 322 | 104
  rSBA-MenA (PI [M36]) | 1238.4 [1126 to 1361.9] | 596.9 [488.5 to 729.3]
  rSBA-MenC (PI [M36]): number analyzed (Participants) | 337 | 109
  rSBA-MenC (PI [M36]) | 870.3 [757.1 to 1000.4] | 1124.8 [812.3 to 1557.6]
  rSBA-MenW-135 (PI [M36]): number analyzed (Participants) | 336 | 105
  rSBA-MenW-135 (PI [M36]) | 2109.2 [1842.5 to 2414.5] | 332.8 [224.4 to 493.8]
  rSBA-MenY (PI [M36]): number analyzed (Participants) | 338 | 108
  rSBA-MenY (PI [M36]) | 2567.3 [2288.6 to 2879.8] | 848 [682.6 to 1053.5]

15. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: At Year 4
Population: The analysis was performed on the ATP cohort for persistence Year 4, which included all evaluable subjects who received the vaccine during the vaccination phase, without a previous dose of meningococcal serogroup A, C, W-135, or Y vaccines and who had available results for at least one tested antigen at the Year 4 time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 312 | 107
Participants
  rSBA-MenA (PI [M48]) ≥ 1:8 | 270 | 79
  rSBA-MenA (PI [M48]) ≥ 1:128 | 245 | 66
  rSBA-MenC (PI [M48]) ≥ 1:8 | 276 | 90
  rSBA-MenC (PI [M48]) ≥ 1:128 | 254 | 79
  rSBA-MenW-135 (PI [M48]) ≥ 1:8 | 231 | 27
  rSBA-MenW-135 (PI [M48]) ≥ 1:128 | 214 | 22
  rSBA-MenY (PI [M48]) ≥ 1:8: number analyzed (Participants) | 309 | 107
  rSBA-MenY (PI [M48]) ≥ 1:8 | 256 | 47
  rSBA-MenY (PI [M48]) ≥ 1:128: number analyzed (Participants) | 309 | 107
  rSBA-MenY (PI [M48]) ≥ 1:128 | 243 | 37

16. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as Geometric Mean Titers (GMTs).
Time Frame: At Year 4
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 312 | 109
Titer
  rSBA-MenA (PI [M48]): number analyzed (Participants) | 312 | 107
  rSBA-MenA (PI [M48]) | 278.6 [219.7 to 353.2] | 105.4 [67.6 to 164.4]
  rSBA-MenC (PI [M48]): number analyzed (Participants) | 312 | 107
  rSBA-MenC (PI [M48]) | 273.6 [220.6 to 339.4] | 315 [196.8 to 504.1]
  rSBA-MenW-135 (PI [M48]): number analyzed (Participants) | 312 | 107
  rSBA-MenW-135 (PI [M48]) | 175.1 [131.5 to 233] | 11.3 [7.8 to 16.3]
  rSBA-MenY (PI [M48]): number analyzed (Participants) | 309 | 107
  rSBA-MenY (PI [M48]) | 350.5 [268.9 to 456.7] | 26 [16.6 to 40.7]

17. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: At Year 5
Population: The analysis was performed on the ATP cohort for persistence Year 5, which included all evaluable subjects who received the vaccine during the vaccination phase, without a previous dose of meningococcal serogroup A, C, W-135, or Y vaccines and who had available results for at least one tested antigen at the Year 5 time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 51 | 19
Participants
  rSBA-MenA (PI [M60]) ≥ 1:8 | 43 | 11
  rSBA-MenA (PI [M60]) ≥ 1:128 | 39 | 3
  rSBA-MenC (PI [M60]) ≥ 1:8: number analyzed (Participants) | 51 | 18
  rSBA-MenC (PI [M60]) ≥ 1:8 | 37 | 7
  rSBA-MenC (PI [M60]) ≥ 1:128: number analyzed (Participants) | 51 | 18
  rSBA-MenC (PI [M60]) ≥ 1:128 | 28 | 5
  rSBA-MenW-135 (PI [M60]) ≥ 1:8 | 44 | 6
  rSBA-MenW-135 (PI [M60]) ≥ 1:128 | 38 | 6
  rSBA-MenY (PI [M60]) ≥ 1:8 | 47 | 12
  rSBA-MenY (PI [M60]) ≥ 1:128 | 47 | 11

18. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as Geometric Mean Titers (GMTs).
Time Frame: At Year 5
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 51 | 19
Titer
  rSBA-MenA (PI [M60]) | 189.8 [107.7 to 334.6] | 37 [12.6 to 108.7]
  rSBA-MenC (PI [M60]): number analyzed (Participants) | 51 | 18
  rSBA-MenC (PI [M60]) | 78.5 [41.8 to 147.4] | 17.3 [6 to 49.7]
  rSBA-MenW-135 (PI [M60]) | 281.6 [145.9 to 543.2] | 15.4 [5.7 to 41.9]
  rSBA-MenY (PI [M60]) | 769.7 [438.6 to 1351] | 74.1 [21.9 to 250.3]

19. Secondary Outcome: Number of Subjects With Anti-PS Antibodies
Description: The cut-off value for the anti-PS concentration was greater than or equal to (≥) 0.3 μg/mL and ≥ 2.0 μg/mL.
Time Frame: At Year 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 354 | 117
Participants
  Anti-PSA (PI [M12]) ≥ 0.3 μg/mL: number analyzed (Participants) | 352 | 116
  Anti-PSA (PI [M12]) ≥ 0.3 μg/mL | 351 | 116
  Anti-PSA (PI [M12]) ≥ 2.0 μg/mL: number analyzed (Participants) | 352 | 116
  Anti-PSA (PI [M12]) ≥ 2.0 μg/mL | 332 | 115
  Anti-PSC (PI [M12]) ≥ 0.3 μg/mL | 349 | 117
  Anti-PSC (PI [M12]) ≥ 2.0 μg/mL | 262 | 113
  Anti-PSW-135 (PI [M12]) ≥ 0.3 μg/mL: number analyzed (Participants) | 348 | 115
  Anti-PSW-135 (PI [M12]) ≥ 0.3 μg/mL | 342 | 112
  Anti-PSW-135 (PI [M12]) ≥ 2.0 μg/mL: number analyzed (Participants) | 348 | 115
  Anti-PSW-135 (PI [M12]) ≥ 2.0 μg/mL | 264 | 102
  Anti-PSY (PI [M12]) ≥ 0.3 μg/mL: number analyzed (Participants) | 354 | 116
  Anti-PSY (PI [M12]) ≥ 0.3 μg/mL | 350 | 116
  Anti-PSY (PI [M12]) ≥ 2.0 μg/mL: number analyzed (Participants) | 354 | 116
  Anti-PSY (PI [M12]) ≥ 2.0 μg/mL | 289 | 110

20. Secondary Outcome: Concentration of Anti-PS Antibodies
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) and measured in µg/mL.
Time Frame: At Year 1
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 354 | 117
μg/mL
  Anti-PSA (PI [M12]): number analyzed (Participants) | 352 | 116
  Anti-PSA (PI [M12]) | 23.25 [19.78 to 27.32] | 31.72 [24.77 to 40.63]
  Anti-PSC (PI [M12]) | 4.67 [4.08 to 5.33] | 24.53 [19.92 to 30.2]
  Anti-PSW-135 (PI [M12]): number analyzed (Participants) | 348 | 115
  Anti-PSW-135 (PI [M12]) | 5.48 [4.68 to 6.4] | 10.39 [7.8 to 13.85]
  Anti-PSY (PI [M12]): number analyzed (Participants) | 354 | 116
  Anti-PSY (PI [M12]) | 6.68 [5.69 to 7.85] | 16.7 [12.9 to 21.6]

21. Secondary Outcome: Number of Subjects With Anti-PS Antibodies
Description: The cut-off value for the anti-PS concentration was greater than or equal to (≥) 0.3 μg/mL and ≥ 2.0 μg/mL.
Time Frame: At Year 2
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 343 | 112
Participants
  Anti-PSA (PI [M24]) ≥ 0.3 μg/mL: number analyzed (Participants) | 336 | 105
  Anti-PSA (PI [M24]) ≥ 0.3 μg/mL | 335 | 105
  Anti-PSA (PI [M24]) ≥ 2.0 μg/mL: number analyzed (Participants) | 336 | 105
  Anti-PSA (PI [M24]) ≥ 2.0 μg/mL | 301 | 103
  Anti-PSC (PI [M24]) ≥ 0.3 μg/mL: number analyzed (Participants) | 340 | 111
  Anti-PSC (PI [M24]) ≥ 0.3 μg/mL | 323 | 111
  Anti-PSC (PI [M24]) ≥ 2.0 μg/mL: number analyzed (Participants) | 340 | 111
  Anti-PSC (PI [M24]) ≥ 2.0 μg/mL | 196 | 107
  Anti-PSW-135 (PI [M24]) ≥ 0.3 μg/mL: number analyzed (Participants) | 336 | 110
  Anti-PSW-135 (PI [M24]) ≥ 0.3 μg/mL | 316 | 108
  Anti-PSW-135 (PI [M24]) ≥ 2.0 μg/mL: number analyzed (Participants) | 336 | 110
  Anti-PSW-135 (PI [M24]) ≥ 2.0 μg/mL | 226 | 93
  Anti-PSY (PI [M24]) ≥ 0.3 μg/mL | 325 | 110
  Anti-PSY (PI [M24]) ≥ 2.0 μg/mL | 237 | 97

22. Secondary Outcome: Concentration of Anti-PS Antibodies
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) and measured in µg/mL.
Time Frame: At Year 2
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 343 | 112
μg/mL
  Anti-PSA (PI [M24]): number analyzed (Participants) | 336 | 105
  Anti-PSA (PI [M24]) | 15.15 [12.76 to 17.98] | 24.85 [19.08 to 32.36]
  Anti-PSC (PI [M24]): number analyzed (Participants) | 340 | 111
  Anti-PSC (PI [M24]) | 2.62 [2.27 to 3.03] | 15.74 [12.56 to 19.72]
  Anti-PSW-135 (PI [M24]): number analyzed (Participants) | 336 | 110
  Anti-PSW-135 (PI [M24]) | 3.51 [2.98 to 4.15] | 6.76 [5.08 to 9.01]
  Anti-PSY (PI [M24]) | 4.44 [3.73 to 5.3] | 11.11 [8.39 to 14.71]

23. Secondary Outcome: Number of Subjects With Anti-PS Antibodies
Description: as for outcome 5
Time Frame: At Year 3
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 331 | 110
Participants
  Anti-PSA (PI [M36]) ≥ 0.3 μg/mL: number analyzed (Participants) | 330 | 109
  Anti-PSA (PI [M36]) ≥ 0.3 μg/mL | 328 | 109
  Anti-PSA (PI [M36]) ≥ 2.0 μg/mL: number analyzed (Participants) | 330 | 109
  Anti-PSA (PI [M36]) ≥ 2.0 μg/mL | 300 | 108
  Anti-PSC (PI [M36]) ≥ 0.3 μg/mL | 318 | 110
  Anti-PSC (PI [M36]) ≥ 2.0 μg/mL | 200 | 106
  Anti-PSW-135 (PI [M36]) ≥ 0.3 μg/mL: number analyzed (Participants) | 328 | 108
  Anti-PSW-135 (PI [M36]) ≥ 0.3 μg/mL | 303 | 105
  Anti-PSW-135 (PI [M36]) ≥ 2.0 μg/mL: number analyzed (Participants) | 328 | 108
  Anti-PSW-135 (PI [M36]) ≥ 2.0 μg/mL | 204 | 87
  Anti-PSY (PI [M36]) ≥ 0.3 μg/mL: number analyzed (Participants) | 323 | 110
  Anti-PSY (PI [M36]) ≥ 0.3 μg/mL | 299 | 108
  Anti-PSY (PI [M36]) ≥ 2.0 μg/mL: number analyzed (Participants) | 323 | 110
  Anti-PSY (PI [M36]) ≥ 2.0 μg/mL | 213 | 92

24. Secondary Outcome: Concentration of Anti-PS Antibodies
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) and measured in µg/mL.
Time Frame: At Year 3
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 331 | 110
μg/mL
  Anti-PSA (PI [M36]): number analyzed (Participants) | 330 | 109
  Anti-PSA (PI [M36]) | 12.5 [10.7 to 14.6] | 19.8 [15.7 to 24.9]
  Anti-PSC (PI [M36]) | 2.7 [2.3 to 3] | 13.9 [11.2 to 17.2]
  Anti-PSW-135 (PI [M36]): number analyzed (Participants) | 328 | 108
  Anti-PSW-135 (PI [M36]) | 2.9 [2.5 to 3.4] | 5.5 [4.2 to 7.2]
  Anti-PSY (PI [M36]): number analyzed (Participants) | 323 | 110
  Anti-PSY (PI [M36]) | 3.8 [3.2 to 4.5] | 8.2 [6.2 to 10.8]

25. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 Pain = pain that prevented normal activity. Grade 3 Redness/Swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 370 | 124
Participants
  Any Pain | 143 | 40
  Grade 3 Pain | 7 | 1
  Any Redness | 57 | 8
  Grade 3 Redness | 1 | 0
  Any Swelling | 42 | 4
  Grade 3 Swelling | 1 | 0

26. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms and headache. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects from whom data were available and who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 371 | 125
Participants
  Any Fatigue | 55 | 13
  Grade 3 Fatigue | 1 | 0
  Related Fatigue | 35 | 8
  ≥ 37.5 ˚C Fever | 16 | 4
  >39.5 ˚C Fever | 0 | 0
  Related Fever | 10 | 2
  Any Gastrointestinal | 13 | 5
  Grade 3 Gastrointestinal | 2 | 0
  Related Gastrointestinal | 6 | 0
  Any Headache | 65 | 15
  Grade 3 Headache | 3 | 0
  Related Headache | 41 | 8

27. Secondary Outcome: Number of Subjects With New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Day 0 up to 6 Months after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 374 | 126
Participants | 1 | 0

28. Secondary Outcome: Number of Subjects With Rash
Time Frame: From Day 0 up to 6 Months after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 374 | 126
Participants | 0 | 1

29. Secondary Outcome: Number of Subjects With AEs Resulting in Emergency Rooms Visits
Time Frame: From Day 0 up to 6 Months after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 374 | 126
Participants | 0 | 0

30. Secondary Outcome: Number of Subjects With Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Up to 31 Days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 374 | 126
Participants | 18 | 8

31. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to 6 Months after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 374 | 126
Participants | 1 | 0

32. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 31
Time Frame: At Year 1, Year 2, Year 3, Year 4 and Year 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 364 | 121
Participants
  Any (SAE)s Year 1 | 0 | 0
  Any (SAE)s Year 2 | 0 | 0
  Any (SAE)s Year 3 | 0 | 0
  Any (SAE)s Year 4 | 0 | 0
  Any (SAE)s Year 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Occurrence of solicited local and general symptoms: during the 4-day (Days 0-3) post vaccination period; Occurrence of unsolicited AE(s): up to 31 days after vaccination; Occurrence of SAE(s): from Day 0 up to 6 months after vaccination.
Description: The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Arm/Group | Nimenrix Group | Mencevax Group
All-Cause Mortality (participants affected / at risk) | 0/374 | 0/126
Serious Adverse Events (participants affected / at risk) | 1/374 | 0/126
Other Adverse Events (participants affected / at risk) | 186/374 | 53/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Group (N=374) | Mencevax Group (N=126)
Mental disorder (Psychiatric disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix Group (N=374) | Mencevax Group (N=126)
Any Pain (General disorders) | 143/370 | 40/124 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Any Redness (General disorders) | 57/370 | 8/124 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Any Swelling (General disorders) | 42/370 | 4/124 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Any Fatigue (General disorders) | 55/371 | 13/125 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Any Headache (General disorders) | 65/371 | 15/125 — This solicited general symptom was only collected from subjects with their symptom sheets completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.